CLINICAL TRIAL: NCT05603338
Title: Naturally Banded Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, assistant professor of general surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fac.med 22.33
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSG (Active Comparator): just laparoscopic sleeve gastrectomy without banding
  Interventions: Procedure: LSG
- LSG with omental band (Experimental): laparoscopic sleeve gastrectomy with omental banding
  Interventions: Procedure: LSG with omental band

INTERVENTIONS:
Procedure: LSG with omental band — LSG with omental band
  Arms: LSG with omental band
Procedure: LSG — just to do sleeve gastrectomy
  Arms: LSG

SUMMARY:
the idea is to use an omental flap or round ligament as a natural band in stead of synesthetic band in bariatric procedures, mainly gastric sleeve

DETAILED DESCRIPTION:
the idea is to use an omental flap or round ligament as a natural band in stead of synesthetic band in bariatric procedures, mainly gastric sleeve

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* patients fit for laparoscopic surgery
* give approval to share in the study
* previous restrictive bariatric procedure

Exclusion Criteria:

* patients unfit for surgery
* patients aged less than 18 and older than 60
* patient with previous upper abdominal surgery either for obesity or other diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
the effect on weight loss | 12 months
  the effect on weight loss determined by percentage of excess weight loss, percentage of total weight loss and change of BMI
the size of gastric pouch at one year | 12 months
  the size of gastric pouch after sleeve gastrectomy in cc at one year using gastric volumetric study

SECONDARY OUTCOMES:
the effect on comorbidities | 12 monthts
  change in comorbidities including diabetes by change in hemoglobin C level, hypertension by measuring arterial blood pressure using sphygmomanometer
operative time | 6 hours
  operative time in minutes from skin incision to skin closure
the incidences of complications | 12 monthss
  the incidences of complications including early complication like leak and bleeding and late complications like stricture diagnosed by vomiting's and imaging and GERD dignosed by symptoms and endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university hospital, Minya, Egypt